CLINICAL TRIAL: NCT04952350
Title: Atorvastatin in Hospitalized COVID-19 Patients: A Randomized, Double-blinded, Placebo-Controlled, Clinical Trial
Brief Title: Atorvastatin for Reduction of 28-day Mortality in COVID-19: RCT
Acronym: COVID-STAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R.21.04.1300.R1
Record Dates: First submitted 2021-07-01; First posted 2021-07-07 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Covid19; SARS-CoV2 Infection; COVID-19 Pneumonia
Keywords: Atorvastatin; randomized clinical trial
MeSH Terms: conditions — COVID-19 | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, caregivers, data collectors, and data analysts will be blinded for the study group. The Delta Pharma company (Egypt) will provide the atorvastatin and a similar placebo. The company will not participate in any step of the study including participant recruitment, data collection, data analysis, or results reporting. The company will prepare a similar package of drug and placebo (labeled as A and B). Even the pharmacist involved in treatment allocation will not know what is the treatment group, just A or B. For emergency unmasking, one of the directors of the COVID19 research council, who will not participate in the study, will know the true labels and the randomization table.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Active Comparator): All patients will be randomized to receive atorvastatin 40 mg once daily orally for a maximum of 28 days. All patients will receive the standard of care according to recent local hospital protocol. Antiviral treatment will be allowed and will be reported.
  Administration in unconscious or ventilated patients: The patients will receive the drug (divided into 4 quadrants) through a nasogastric tube.
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet
- Control (Placebo Comparator): All patients will be randomized to receive the placebo once daily orally for a maximum of 28 days. All patients will receive the standard of care according to recent local hospital protocol. Antiviral treatment will be allowed and will be reported.
  Administration in unconscious or ventilated patients: The patients will receive the drug through a nasogastric tube.
  Placebo will resemble the original drug as regards the drug package, the tablet color, consistency, and size.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet — Patients will receive Atorvastatin 40 mg orally within 24 hrs after hospital admission after evaluation of the clinical and laboratory inclusion criteria.
  Other Names: 134523-00-5; ATORVASTATIN CALCIUM; Lipitor
  Arms: Atorvastatin
Other: Placebo — A formulary similar to the drug tablets and labels but without the active ingredients (Atorvastatin).
  Arms: Control

SUMMARY:
This randomized placebo-controlled double-blinded clinical trial aims to test the efficacy of administering atorvastatin 40 mg to hospitalized COVID-19 patients for 28 days on the all-cause 28-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* We will include adult patients (≥18 years old) with severe and critical COVID19 admitted to the COVID19 Mansoura University isolation hospital. We will include patients who are PCR-confirmed, clinically or radiologically diagnosed with COVID19.

Cases are defined as severe or critical according to the WHO definition (19); where critical cases have ARDS, or sepsis, septic shock or pulmonary embolism, acute coronary syndrome, or acute stroke, while severe cases have the clinical signs of severe pneumonia and SpO2 <90% on room air, or RR <30 breaths/min without any critical criteria.

Exclusion Criteria:

* chronic statin use, serum creatine kinase (sr CK) > 5 times the upper limit of normal (ULN), serum transaminases > 5 times ULN, acute hepatic failure, chronic liver disease (Child-Pugh Classification C), history of rhabdomyolysis or myopathies, severe renal impairment not receiving renal replacement therapy (estimated Cr cl< 30 ml\min ), pregnant and lactating women, patients who are expected to die within 48 hours, or patients on chronic colchicine, cyclosporines, or ritonavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days after randomization
  all-cause mortality
mortality | 6 months after randomization
  all-cause mortality

SECONDARY OUTCOMES:
incidence of invasive mechanical ventilation (IMV) | 28 days or primary hospital stay
  incidence
duration of invasive mechanical ventilation (IMV) | 28 days or primary hospital stay
  duration in days
Time to clinical improvement | 28 days or primary hospital stay
  2 points reduction in the WHO disease ordinal progression scale or discharge, whatever happens first.
serious adverse effects | 28 days after start of the drug
  any event that leads to discontinuation of the drug
Intensive Care length of stay | 28 days or primary hospital stay
  duration in days
acute kidney injury | 28 days or primary hospital stay
  Increase in Scr by >/ 0.3 mg/ dl in 48 hr or Increase in Scr by >/ 50% in 7 days or Oliguria for >/ 6 hours.
status at hospital discharge | through study completion, an average of 9 months
  dead or alive
Hospital length of stay | through study completion, an average of 9 months
  Length of hospital stay in days

OTHER OUTCOMES:
C-Reactive Protein | on days 3, 7, 14, and 28 after randomization/ if still hospitalized
  as inflammatory marker
Sequential Organ Failure Assessment scale | on days 3, 7, 14, and 28 after randomization/ if still hospitalized
  SOFA scale
COVID Disease progression score | on days 3, 7, 14, and 28 after randomization/ if still hospitalized
  according to the January 2021 WHO update

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Study Director — Mansoura University - Faculty of Medicine
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We will make the anonymous individual data available at reasonable request after publication. Patient confidentiality will be kept safe.
Time Frame: will be updtaed shortly
Access Criteria: will be updated shortly

REFERENCES:
- [Derived] Eltahan NH, Elsawy NH, Abdelaaty KM, Elhamaky AS, Hassan AH, Emara MM. Atorvastatin for reduction of 28-day mortality in severe and critical COVID-19 patients: a randomized controlled trial. Respir Res. 2024 Feb 22;25(1):97. doi: 10.1186/s12931-024-02732-2. PMID 38389078
- [Derived] Emara MM, Elsawy NH, Abdelaaty KM, Elhamaky AS, Eltahan NH. Atorvastatin for reduction of 28-day mortality in hospitalized COVID-19 patients: study protocol for a randomized, double-blinded, placebo-controlled, clinical trial. Trials. 2022 Aug 8;23(1):636. doi: 10.1186/s13063-022-06619-9. PMID 35941669